CLINICAL TRIAL: NCT06054425
Title: A Phase 1 Pharmacokinetic Comparability Study in Healthy Subjects to Evaluate the Relative Bioavailability of Risankizumab in Vials Manufactured by Two Different Processes
Brief Title: A Study to Compare the Bioavailability of Intravenously Infused Risankizumab Manufactured by Two Different Processes in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M24-696
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers
Keywords: Risankizumab
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Participants will receive risankizumab manufactured with using the current process (CMC2).
  Interventions: Drug: Risankizumab
- Arm 2 (Active Comparator): Participants will receive risankizumab manufactured with using the new process (CMC3).
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Infusion; intravenous

SUMMARY:
The objective of this study is to assess the bioavailability of risankizumab liquid vial manufactured with the new process (CMC3) relative to the current process (CMC2).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) >= 18.0 to <= 32.0 kg/m2 after rounding to the tenths decimal at the time of screening and upon initial confinement.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).
* Body weight less than 100.00 kg at Screening and upon initial confinement.

Exclusion Criteria:

* History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.
* Previous exposure to any anti-interleukin (IL)-12/23 or anti-IL-23 treatment for at least one year prior to Screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | Up to Day 131
  Cmax will be assessed.
Time to Cmax (Tmax) | Up to Day 131
  Tmax will be assessed.
Apparent Terminal Phase Elimination Rate Constant (β) | Up to Day 131
  Apparent terminal phase elimination rate constant (β) will be assessed.
Terminal Phase Elimination Half-life (t1/2) | Up to Day 131
  Terminal phase elimination half-life (t1/2) will be assessed.
Area Under the Concentration-time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUC0-t) | Up to Day 131
  AUC0-t will be assessed.
AUC from Time 0 to Infinity (AUC0-inf) | Up to Day 131
  AUC0-inf will be assessed.
Number of Participants with Adverse Events (AEs) | Baseline to Day 141
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (3):
- United States (3):
  - Anaheim Clinical Trials LLC /ID# 260740, Anaheim, California
  - Clinical Pharmacology of Miami /ID# 260800, Miami, Florida
  - Acpru /Id# 260864, Grayslake, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-696